CLINICAL TRIAL: NCT01021202
Title: Early vs. Late Percutaneous Dilation Tracheostomy in Mechanically Ventilated Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Timing of Dilation Tracheostomy in Mechanically Ventilated Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unexpectedly slow recruitment
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KIM-PV3278/UKE
Record Dates: First submitted 2009-10-06; First posted 2009-11-26 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: tracheostomy; tracheotomy; dilational; dilatative; critical care; intensive care; COPD; chronic obstructive pulmonary disease; lung disease; pneumonia; prospective study; questionnaire; quality of life; outcome; mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early tracheostomy (Experimental): Percutaneous dilation tracheostomy < 72h on mechanical ventilation
  Interventions: Procedure: Percutaneous dilation tracheostomy
- Late tracheostomy (Experimental): Percutaneous dilation tracheostomy > 10 days on mechanical ventilation
  Interventions: Procedure: Percutaneous dilation tracheostomy

INTERVENTIONS:
Procedure: Percutaneous dilation tracheostomy — Percutaneous dilation tracheostomy using Ciaglia blue rhino system (Cook medical, Limerick, IRELAND). Tracheostomy is conducted by two experienced physicians with (video-)bronchoscopic control and continuous monitoring of ECG, blood pressure, pulse and peripheral oxygen saturation.

SUMMARY:
The purpose of this study is:

* to evaluate the optimal time-point for percutaneous dilation tracheostomy in COPD patients in terms of duration on mechanical ventilation, length of stay on ICU and mortality;
* to evaluate the rate of infections and infectious complications of tracheostomized COPD patients;
* to evaluate the spectrum of pathogens in tracheostomized and intubated COPD patients;
* to evaluate the amount of sedatives used in mechanically ventilated COPD patients;
* to assess the quality of life in COPD patients tracheostomized after 3 or after 10 days.

DETAILED DESCRIPTION:
Screening of patients following inclusion and exclusion criteria on all units of the Department of Critical Care will occur on a daily basis.

Randomization will be performed by blocks of sealed envelopes containing random numbers which are deposited at a central space within the Department of Critical Care Medicine. Randomization is performed as permuted block randomization.

Collection of baseline parameters (last/current lung function test, last/current 6-min walk test, cardiac stress test - if accessible) If not accessible, current lung function test results (at least FEV1 and FVC) are requested from the patient's general physician or pulmonologist to determine GOLD stage.

Patients randomized into the (early tracheostomy) study group, will undergo tracheostomy at the next possible opportunity but not later than 72 h after initiation of invasive ventilation. Patients of the control group will be invasively ventilated at least until Day 10.

Before tracheostomy a complete endoscopic inspection of the bronchial system will be performed routinely. Bronchoalveolar lavage fluid (BALF) will be obtained from sites of pulmonary infiltrations. In case of no radiographically or bronchoscopic detectable infiltrations BALF will be drawn from the Middle Lobe.

Primary and secondary endpoints will be analyzed at given time-points.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (GOLD stage III or IV)
* Suspected long-time invasive mechanical ventilation due to ARF (> 10 days)
* Informed consent of the patient or legal guardian

Exclusion Criteria:

* Severe neurological failure (such as stroke, cerebral haemorrhage etc.)
* Immunosuppressant therapy (with the exception of steroid therapy)
* Major risk of bleeding
* Intubation > 72 h
* Contraindication for dilation tracheotomy
* Impossibility of intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cumulative duration of mechanical ventilation (in days) | Day 1 - 28
  Cumulative duration of mechanical ventilation (in days)

SECONDARY OUTCOMES:
All-cause mortality | Day 28, 90 and end of ICU stay
  All-cause mortality
Length of stay on ICU / hospital | end of ICU / hospital stay
  Length of stay on ICU / hospital
Infections (Ventilator-associated pneumonia, spectrum of pathogens in BALF, infectious complications) | Day 1 - 28
  Infections (Ventilator-associated pneumonia, spectrum of pathogens in BALF, infectious complications)
Cumulative use of sedatives | Day 1 - 28
  Cumulative use of sedatives
Quality of Life - Questionnaire | discharge from ICU, day 28 and day 90
  Quality of Life - Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, Principal Investigator — Department of Critical Care Medicine, University Medical Center Hamburg - Eppendorf
Locations (1):
- Universitätsklinikum Hamburg - Eppendorf (University Medical Center Hamburg-Eppendorf), Hamburg, Germany